CLINICAL TRIAL: NCT06384833
Title: Combination of Vitamin C and N-Acetylcysteine to Improve Functional Outcome After Rotator Cuff Repair: A Triple-blinded, Randomized Controlled Trial
Brief Title: Combination of Vitamin C and N-Acetylcysteine to Improve Functional Outcome After Rotator Cuff Repair
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rama
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tears
Keywords: Ascorbic acid; Acetylcysteine; Rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ascorbic Acid; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ascorbic Acid and N-acetylcysteine (Experimental): Vitamin C 500 mg IV q4h for 4 doses PO d0 N-acetylcysteine 600mg 1 tab PO OD for 45 days Vitamin C 100mg 5 tab PO BID for 45 days
  Interventions: Drug: Ascorbic acid; Drug: N-acetyl cysteine
- Placebo (Placebo Comparator): Placebo of vitamin C (0.9%NaCl) 100 ml IV q4h for 4 doses PO day0 Placebo of N-acetylcysteine 1 tab PO OD for 45 days Placebo of Vitamin C 5 tab PO BID for 45 days
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Ascorbic acid — Vitamin C (solution) 500 mg IV q4h for 4 doses PO d0 Vitamin C (tablet) 100mg 5 tab PO BID for 45 days
  Other Names: Vitamin C
  Arms: Ascorbic Acid and N-acetylcysteine
Drug: N-acetyl cysteine — NAC (effervescent) 600mg 1 tab PO OD for 45 days
  Other Names: NAC
  Arms: Ascorbic Acid and N-acetylcysteine
Other: placebo — pharmacologically inactive substance
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if vitamin C and N-acetylcysteine work to improve shoulder functional score after rotator cuff repair. It will also learn about the safety of vitamin C and N-acetylcysteine. The main questions it aims to answer are:

Do vitamin C and N-acetylcysteine improve the shoulder functional score of participants? Do vitamin C and N-acetylcysteine improve healing of rotator tendon? Researchers will compare vitamin C and N-acetylcysteine to a placebo (a look-alike substance that contains no drug) to see if vitamin C and N-acetylcysteine works to improve shoulder functional score after rotator cuff repair.

Participants will:

Take vitamin C and N-acetylcysteine or a placebo every day for 45 days. Visit the OPD three times at 2 week, 6 month and 12 month after surgery for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* All patient who undergone arthroscopic primary rotator cuff complete repair.
* Clinical history and symptom consistent with rotator cuff tear.
* MRI confirmation of rotator cuff tear.

Exclusion Criteria:

* Non-reparable or partial rotator cuff repair.
* High grade fatty degeneration of the rotator cuff (Goutallier III, IV)
* At least one torn tendon with retraction to the glenoid (stage 3 of Patte classification)
* Rotator cuff retear.
* Isolated subscapularis tear.
* Patient who loss follow up.
* Patent who cannot respond questionnaire.
* Patient who allergy to vitamin C or N-acetylcysteine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
ASES score | 6 months after surgery
  American Shoulder and Elbow Surgeons (ASES) Shoulder Score

SECONDARY OUTCOMES:
UCLA shoulder scale | 6 months after surgery
  The University of California-Los Angeles (UCLA) shoulder scale
WORC index | 6 months after surgery
  Western Ontario Rotator Cuff Index
Tendon healing at 6 months postoperatively | 6 months after surgery
  Sugaya ultrasound classification

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uehara H, Itoigawa Y, Morikawa D, Koga A, Tsurukami H, Maruyama Y, Ishijima M. The Effect of Vitamin C and N-Acetylcysteine on Tendon-to-Bone Healing in a Rodent Model of Rotator Cuff Repair. Am J Sports Med. 2023 May;51(6):1596-1607. doi: 10.1177/03635465231160772. Epub 2023 Apr 5. PMID 37017249
- [Background] Gilat R, Atoun E, Cohen O, Tsvieli O, Rath E, Lakstein D, Levy O. Recurrent rotator cuff tear: is ultrasound imaging reliable? J Shoulder Elbow Surg. 2018 Jul;27(7):1263-1267. doi: 10.1016/j.jse.2017.12.017. Epub 2018 Feb 3. PMID 29398398
- [Result] Martel M, Laumonerie P, Girard M, Dauzere F, Mansat P, Bonnevialle N. Does vitamin C supplementation improve rotator cuff healing? A preliminary study. Eur J Orthop Surg Traumatol. 2022 Jan;32(1):63-70. doi: 10.1007/s00590-021-02926-0. Epub 2021 Mar 16. PMID 33725178